CLINICAL TRIAL: NCT04031963
Title: Novel Biophotonics Methodology for Colon Cancer Screening
Acronym: BRP
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Collaborators: Northwestern University (Other); University of Chicago (Other); Indiana University (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: R01CA128641 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Colon Cancer
Keywords: Novel Biophotonic Methodology for Colon Cancer Screening.
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Those with colon cancer and with adenomatous polyp and those without a previously mentioned condition.

SUMMARY:
This is a proposal to establish a Bioengineering Research Partnership (BRP). The major objective of the BRP is to refine and provide comprehensive, definitive multi-center validation of these novel methodologies for colorectal cancer (CRC) screening, thus providing a quantum leap in population screening.

DETAILED DESCRIPTION:
Background and Significance highlights the impracticality to provide total colonic evaluation for the entire population. Risk-stratification via exploitation of the "field effect" is an attractive approach. However, all existing methodologies (e.g FOBT, fecal DNA, flexible sigmoidoscopy) are clearly suboptimal underscoring the need for novel tools for identifying the field effect.

1) We have developed ELF/LEBS for depth-selective (from ~30 to hundreds of microns) spectroscopic assessment of living tissue. 2) We tested these novel techniques in two animal models of CRC (the AOM-treated rat and MIN-mouse) and in human subjects (n=190). We demonstrated that ELF/LEBS has the potential to detect precancerous changes in the colon at a time point that precedes the formation of adenomas and other histological/molecular markers of CRC. 3) We demonstrated that rectal ELF/LEBS can detect field effect alterations in histologically normal rectal tissue changes due to the presence of adenomas anywhere in the colon. In our pilot studies, the diagnostic accuracy of rectal ELF/LEBS far exceeded any other currently known markers of CRC. Therefore, assaying ELF/LEBS in the rectum has the potential to provide accurate risk-stratification for colon carcinogenesis without the need for bowel preparation and colonoscopy. 4) We have developed prototypes of ELF and LEBS fiber-optics probes for in vivo use.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years old or older and is having a colonoscopy procedure.

Exclusion Criteria:

* Concurrent usage of anticoagulation or blood thinner medication within the last 7 days that would preclude Hx of Inflammatory Bowel Disease/Colitis/Chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients going under colonoscopy or sigmoidoscopy procedure.
Sampling Method: Probability Sample
Enrollment: 857 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Early cancer changes in the colon | Visit 1, screening colonoscopy
  ELF/LEBS probe used to obtain spectroscopy readings from rectal tissue

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Roy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore Univeristy HealthSystems, Evanston, Illinois, United States